CLINICAL TRIAL: NCT06002022
Title: Local Intervention Trial for the Evaluation of Improvements in Patient-reported Quality of Life and Treatment Satisfaction in BCP as a Result of Flexible Treatment Planning Supported by REBECCA-collected RWD
Brief Title: Evaluation of Improvements in Patient-reported Quality of Life
Acronym: REBECCA-QoL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/005-QoL
Record Dates: First submitted 2023-02-03; First posted 2023-08-21 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Quality of Life; Physical Activity; Sleep Quality; Stress; Pain
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Sleep Initiation and Maintenance Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Control arm: Patients will be treated as usual after the first-line breast cancer treatment. Specifically, this process entails biannual medical evaluation control visits for the first port-treatment year at the Oncology Department, including standardised blood examinations.
  Experimental arm: Additionally, patients will be trained in the use of the REBECCA mobile and online monitoring platform, which will be used longitudinally, with the collection of real-world data within the REBECCA framework. Their supervising health personnel will be given access to the REBECCA patient dashboard, which provides in-depth information about their lifestyle, as well as continuous REBECCA measurements for their online behaviour and self- or companion-reported measures of emotional state and quality of life.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (No Intervention): Patients in the control arm will be treated as usual after the first-line breast cancer treatment. Specifically, in Valencia, this process entails biannual medical evaluation control visits for the first port-treatment year at the Oncology Department, including standardised blood examinations.
  On top of that, patients of this group will be offered 3 supportive consultation sessions, over the phone, with generic advice on desired lifestyle choices (physical activity, dietary habits, sleep habits and social mobility) that will be helpful for managing the ongoing treatment
- Standard treatment + REBECCA (Experimental): Patients will be trained in the use of the complementary monitoring modules of the REBECCA mobile and online monitoring platform, which will be used longitudinally, facilitating the collection of real world data within the REBECCA framework. Their supervising health personnel will be given access to the REBECCA patient dashboard, that provides in-depth information about their lifestyle, as well as continuous REBECCA measurements for their online behaviour and self- or companion-reported measures of emotional state and quality of life.
  Unlike those in the "Standard care" study-arm, 3 phone-based consultation sessions in the first 12 months of treatment visits will be scheduled based on system-predicted eminent life functionality and emotional state deteriorations (and potential decrease in treatment compliance), targeting the just-in-time patient support, aiming at improving treatment acceptance and efficacy
  Interventions: Device: REBECCA system (smartwatch + mobile app use)

INTERVENTIONS:
Device: REBECCA system (smartwatch + mobile app use) — Patients will be trained in the use of the REBECCA system, which will provide in-depth information about their lifestyle (including physical activity levels, dietary habits, sleep quality and social mobility), as well as of their online behaviour (with outcome indicators of anxiety, PTSD and depression development) and self- or companion-reported measures of emotional state and quality of life. Based on the additional information, exploiting the enhanced monitoring capabilities of the REBECCA system, the supervising clinicians will be given the opportunity to continuously evaluate the progress of the patients, allowing them to schedule up to 3 phone-based consultation sessions in the first 12 months of treatment
  Arms: Standard treatment + REBECCA

SUMMARY:
Local intervention trial for the evaluation of improvements in patient-reported Quality of Life and treatment satisfaction, in breast cancer patients (BCP), as a result of flexible treatment planning supported by REBECCA-collected real-world data, in comparison with standard care

DETAILED DESCRIPTION:
Local intervention trial which will evaluate the potential of using real-world patient measurements collected by the REBECCA system for improving the patient-reported quality-of-life, through just-in-time support consultations, during the first 12 months after radiology and/or chemotherapy treatment. The effects of the REBECCA-assisted treatment on QoL, in relation to baseline, will be compared against standard

The use of REBECCA-collected patient information by BCP-supervising health professionals (based on the continuous REBECCA real-world measurements), aims to estimate to which extent it:

- Improves the quality of the provided treatment at 12 months, resulting in an improved QoL, in comparison with standard treatment practice

It will also evaluate that:

* The observed improvements will persist long-term, at least till the point of the 18-month follow-up evaluation
* The observed QoL improvements will be associated with REBECCA's Functional Life Index improvements, as evaluated through the continuous REBECCA real world measurements. This will act as an assessment of the RWD use for safer and more effective post-treatment management of interventions with first line chemo/radiotherapies in breast cancer.
* The observed QoL improvements will be associated with REBECCA's PROM Index improvements, as evaluated through the continuous REBECCA real world measurements.

ELIGIBILITY:
Inclusion Criteria:

* Before patient registration, written informed consent must be given according to national and local regulations.
* Participants have had histologically proven stage I-III breast cancer undergoing endocrine treatment (with or without prior chemotherapy) no more than 12 months prior to randomization.
* Be between 18 and 75 years of age.
* Have increased life expectancy beyond the initial 3 months post-treatment initiation.
* Have the ability to understand protocol, participate in testing and willingness to sign a written informed consent.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Exclusion Criteria:

* Patients that are not willing to sign an informed consent form

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 110 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Resting quality | 18 months follow up since enrolment with a monthly measurement
  Emotional state deterioration from QoL questionnaires of the last 24 hours prior to the measurement.
  Scale scored from 1-5 (1 not rested, 5 very rested)
Stress level | 18 months follow up since enrolment with a monthly measurement
  Emotional state deterioration from QoL questionnaires of the last 24 hours prior to the measurement.
  Scale scored from 1-5 (1 not stressed, 5 very stressed)
Stress level related to illness | 18 months follow up since enrolment with a monthly measurement
  Emotional state deterioration from QoL questionnaires of the last 24 hours prior to the measurement.
  Scale scored from 1-5 (1 not stressed, 5 very stressed)
Pain level of the last 24 hours | 18 months follow up since enrolment with a monthly measurement
  Emotional state deterioration from QoL questionnaires of the last 24 hours prior to the measurement.
  Scale scored from 1-5 (1 not bad, 5 very bad)
Tiredness level of the last 24 hours | 18 months follow up since enrolment with a monthly measurement
  Emotional state deterioration from QoL questionnaires of the last 24 hours prior to the measurement.
  Scale scored from 1-5 (1 not tired, 5 very tired)

SECONDARY OUTCOMES:
Weight | 18 months follow up since enrolment
  Weight measurement (kg) as part of the anthropometric examination
Height | 18 months follow up since enrolment
  Height measurement (cm) as part of the anthropometric examination

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://rebeccaproject.eu/

DOCUMENTS (1):
  • Informed Consent Form (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT06002022/ICF_000.pdf